CLINICAL TRIAL: NCT00898118
Title: Serial Analysis of Chimerism in Patients With Refractory Cytopenia (RC) Transplanted With Reduced Intensity Conditioning (RIC)
Brief Title: Studying Blood Samples in Young Patients With Cytopenia After a Donor Stem Cell Transplant
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: European Working Group of MDS in Childhood (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: EWOG-MDS-SCT RC RIC-06; CDR0000587523 (Registry Identifier: PDQ (Physician Data Query)); EU-20808
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2008-04

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: refractory cytopenia with multilineage dysplasia; childhood myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — Polymerase Chain Reaction; Flow Cytometry

INTERVENTIONS:
Genetic: polymerase chain reaction
Other: flow cytometry
Other: laboratory biomarker analysis
Procedure: allogeneic hematopoietic stem cell transplantation

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at blood samples in young patients with cytopenia after undergoing a donor stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To study hematopoietic chimerism in whole blood and different cell populations (i.e., CD14, CD15, CD 56, CD3, and CD19) as well as in dendritic cells and regulatory T cells after allogeneic hematopoietic stem cell transplantation with reduced intensity conditioning in patients with refractory cytopenia.
* To compare the results of chimerism obtained with standard short tandem nucleotide polymorphism PCR (sensitivity 1%) with those obtained with single nucleotide polymorphisms PCR (sensitivity 0.1- 0.01%).

Secondary

* To evaluate the relationship between mixed chimerism and hematological engraftment, overall survival, and event-free survival.
* To study the impact of mixed chimerism in plasmacytoid dendritic and regulatory T cells on the incidence of acute and chronic graft-versus-host-disease.

OUTLINE: This is a multicenter study.

Peripheral blood is collected from patients and donors prior to hematopoietic stem cell transplantation (HSCT). Patients also undergo blood sample collection on days 30, 60, 100, and 180 after transplantation. Peripheral blood cells are enriched and separated into lineage-specific subpopulations (i.e., CD3, CD14, CD15, CD19, and CD56) which are then divided equally for either DNA isolation via PCR or for flow cytometry. DNA concentrations in pre-HSCT donor and patient samples and in post-HSCT subpopulation samples are determined using quantitative real-time PCR. Samples are also analyzed for quantification of chimerism and detection of genetic markers via short tandem repeats- and sequence nucleotide polymorphism-based chimerism analyses.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with refractory cytopenia

  * Hypocellular bone marrow and normal karyotype
* Underwent stem cell transplantation (SCT) from an HLA identical (8/8) sibling, an HLA identical (10/10) relative, or an HLA identical or single allelic disparate unrelated donor

  * Received a preparative regimen including either thiotepa or fludarabine phosphate
* Concurrently enrolled on EWOG-MDS-2006

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Estimated)
Dates: Start 2007-04; Primary Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients with complete chimerism as measured by standard short tandem nucleotide polymorphism PCR in whole blood and the different cell populations
Number of patients with complete chimerism as measured by single nucleotide polymorphisms PCR in the different cell populations

SECONDARY OUTCOMES:
Number of patients with mixed chimerism and full hematological recovery at day 100
Number of patients with mixed chimerism and acute or chronic graft-versus-host disease

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bader, MD, Principal Investigator — European Working Group of MDS in Childhood
Locations (10):
- St. Anna Children's Hospital, Vienna, Austria
- Ghent University, Ghent, Belgium
- University Hospital Motol, Prague, Czechia
- Aarhus Universitetshospital - Aarhus Sygehus, Aarhus, Denmark
- Germany (2):
  - European Working Group of MDS in Childhood, Freiburg im Breisgau
  - Universitaetskinderklinik - Universitaetsklinikum Freiburg, Freiburg im Breisgau
- IRCCS "Casa Sollievo della Sofferenza", South Giovanni Rotondo, Italy
- Erasmus MC - Sophia Children's Hospital, Rotterdam, Netherlands
- Akademia Medyczna im. Piastow Slaskich, Wroclaw, Poland
- University Children's Hospital, Zurich, Switzerland